CLINICAL TRIAL: NCT00609687
Title: Diagnostic Yield of Vitreous Biopsy in Sarcoid Uveitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00014310
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2008-01

CONDITIONS: Sarcoidosis-associated Ocular Inflammation
Keywords: sarcoidosis; diagnostic vitrectomy; vitreous biopsy; sarcoidosis-associated ocular inflammation
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Other): Patients with suspected sarcoid-related posterior segment inflammation with inconclusive clinical exam findings, ancillary testing, and laboratory results
  Interventions: Procedure: Diagnostic Vitrectomy

INTERVENTIONS:
Procedure: Diagnostic Vitrectomy — Three-port, 20-gauge pars plana vitrectomy instrumentation was utilized. An infusion line was inserted into one sclerotomy and secured to the globe. A second sclerotomy was made, and a fiberoptic light pipe was immediately inserted to minimize vitreous egress. A third sclerotomy was created, and the vitreous cutter was inserted. To obtain an undiluted vitreous sample, the vitreous was cut mechanically with the vitreous cutter, while the assistant surgeon simultaneously manually aspirated the vitreous. After sufficient undiluted sample was obtained, infusion fluid was allowed to enter the eye and a diluted vitreous sample was obtained in a similar manner. The samples were personally carried to the clinical laboratories by the operating surgeon.
  Vitreous fluid analysis was guided by clinical suspicion based on the pre-operative differential diagnosis and the intraoperative posterior segment appearance.

SUMMARY:
The usefulness of diagnostic vitrectomy in patients with suspected sarcoidosis with posterior segment involvement (in whom a diagnosis cannot be determined by conventional methods) has not been well described. We hypothesized that diagnostic vitrectomy would help establish the diagnosis in these challenging cases. Herein, we evaluated the diagnostic yield of vitreous biopsy in patients with suspected sarcoidosis-associated uveitis that affected the posterior segment.This is a retrospective interventional case series. Cases of intermediate, posterior or panuveitis that could not be characterized by clinical examination, ancillary, and laboratory tests were considered for diagnostic pars plana vitrectomy. Retrospective chart review was conducted on consecutive eyes that underwent diagnostic, or diagnostic and therapeutic vitrectomy by a single surgeon from January 1989 to June 2006.

DETAILED DESCRIPTION:
We obtained approval to conduct this non-comparative, interventional, retrospective case series from the Duke University Institutional Review Board. We used an established database of patients with uveitis and the operative reports from a single surgeon (GJJ) to identify all consecutive patients who underwent diagnostic pars plana vitrectomy from January 1989 to June 2006. We excluded patients with acute postoperative or traumatic endophthalmitis from this study. Cases were included if intraocular vitreous specimens were obtained for diagnostic testing. After identifying 150 patients, we reviewed the medical records of these individuals as previously described.

Patient demographic data and clinical history were recorded at the time of initial visit. A complete ophthalmic history and examination were performed by a single examiner (GJJ). The examination included slit-lamp biomicroscopy and dilated fundus examination with indirect ophthalmoscopy. Anterior segment inflammation was graded using the system described by Hogan and colleagues. The system previously described by Nussenblatt et.al. was used to grade vitreous opacity. Fluorescein angiography, optical coherence tomography, and ultrasonography were performed as indicated. A differential diagnosis was compiled for each case, based on clinic findings. Additional laboratory tests were ordered depending on the constellation of clinical history, exam findings, and results of previous ancillary testing. Anti-inflammatory therapy was initiated in an empiric or diagnosis-specific manner, and the clinical response was followed carefully.

Diagnostic vitrectomy was performed on eyes with intermediate, posterior, or panuveitis in which an etiology could not be characterized by clinical examination, laboratory, and/or ancillary testing. In addition, diagnostic vitrectomy was performed on eyes that did not adequately respond to empirical therapy, or those in which intraocular malignancy or infection was suspected. Therapeutic vitrectomy was performed in conjunction with diagnostic vitrectomy when clinically indicated, for example to repair retinal detachment, to remove epiretinal membranes, to decrease vitreous opacity, or to insert an intraocular sustained drug-delivery implant.

In this study, vitreous samples were collected in the operating room using a standardized technique which has been previously reported. Briefly, three-port, 20-gauge pars plana vitrectomy instrumentation was utilized. An infusion line was inserted into one sclerotomy and secured to the globe. A second sclerotomy was made, and a fiberoptic light pipe was immediately inserted to minimize vitreous egress. A third sclerotomy was created, and the vitreous cutter was inserted. To obtain an undiluted vitreous sample, the vitreous was cut mechanically with the vitreous cutter, while the assistant surgeon simultaneously manually aspirated the vitreous. The tip of the vitreous cutter was viewed at all times with the wide-field viewing system during the procedure. After sufficient undiluted sample was obtained, infusion fluid was allowed to enter the eye and a diluted vitreous sample was obtained in a similar manner. The samples were personally carried to the clinical laboratories by the operating surgeon. Vitreous fluid analysis was guided by clinical suspicion based on the pre-operative differential diagnosis and the intraoperative posterior segment appearance. Cytopathology was used to identify granulomatous inflammation or tumor cells. A thin-prep was prepared, processed through a membrane filter apparatus (Millipore Corp, Bedford, MA) and then stained with Papanicolaou stain. Gram stain, KOH preparation and culture were used to diagnose intraocular infection. Where appropriate, instructions were given to the clinical laboratory for specific sample processing (e.g., suspected slow-growing bacterium, such as Propionibacterium acnes or suspected fungal infection). Genomic amplification by polymerase chain reaction (PCR) was performed at the University of Colorado (Boulder, CO), or Texas Children's Hospital (Houston, TX) to test for the presence of Herpes simplex virus, Herpes zoster virus, and cytomegalovirus. PCR was performed for Toxoplasma gondii at the Palo Alto Medical Foundation (Palo Alto, CA) as previously described. Toxocara canis antibody levels were detected by enzyme-linked immunosorbent assay (ELISA) at the Centers for Disease Control and Prevention (Atlanta, GA). For Toxoplasma gondii and Toxocara canis, simultaneous serum samples were also collected and sent to the respective laboratories.

The final diagnosis was based upon the results of the directed diagnostic testing of the vitreous sample. A positive diagnostic vitrectomy result was based upon the identification of a specific etiologic agent through the testing modalities previously described. Sarcoidosis is a diagnosis of exclusion without a known etiologic agent. There are no definitive laboratory tests that unequivocally confirm a diagnosis of sarcoid. Therefore, a diagnostic specimen was deemed positive for sarcoid-related inflammation if the following criteria were satisfied: 1) if all other vitreous testing was negative 2) if the clinical features were such that sarcoidosis was included in the differential diagnosis based on pre-operative clinical appearance, and 3) if the cytopathology specimen was consistent with a pattern of sarcoid-related inflammation such as non-caseating granuloma formation, as established by the cytopathologist.

ELIGIBILITY:
Inclusion Criteria:

* Cases were included if intraocular vitreous specimens were obtained for diagnostic testing.

Exclusion Criteria:

* Patients with acute postoperative or traumatic endophthalmitis from this study were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To determine the diagnostic yield of vitreous biopsy in patients with suspected sarcoid uveitis | January 1989 to June 2006

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J Jaffe, MD, Principal Investigator — Duke University Eye Center
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Mruthyunjaya P, Jumper JM, McCallum R, Patel DJ, Cox TA, Jaffe GJ. Diagnostic yield of vitrectomy in eyes with suspected posterior segment infection or malignancy. Ophthalmology. 2002 Jun;109(6):1123-9. doi: 10.1016/s0161-6420(02)01033-3. PMID 12045054
- [Derived] Scott AW, Mruthyunjaya P, McCallum RM, Jaffe GJ. Diagnostic yield of vitreous biopsy in presumed sarcoidosis-related posterior segment inflammation. Graefes Arch Clin Exp Ophthalmol. 2012 Sep;250(9):1379-85. doi: 10.1007/s00417-012-1993-9. Epub 2012 Mar 21. PMID 22434211